CLINICAL TRIAL: NCT06458231
Title: Determining the Prevalence of Primary and Secondary Central Line Associated Blood Stream Infection (CLABSI) at the Tertiary Care Hospital
Acronym: Microbiology
Status: Recruiting | Type: Observational
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Other Study IDs: Micro
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI)
Keywords: CLABSI, Primary B.I., Secondary B.I.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No of Positive CLABSI: No of +ve CLABSI in different types of cases,
  Interventions: Device: Blood Catheters
- Primary Blood stream infection: Participant with blood stream infection not related to other other infection in the body
  Interventions: Device: Blood Catheters
- Secondary Blood stream infection: Blood stream infection occur as a complication to infection in other parts of the body
  Interventions: Device: Blood Catheters
- Blood Prevalence of types microorg.: % and Prevalence of different microorg causing Blood stream infection

INTERVENTIONS:
Device: Blood Catheters — Central line as a predisposing factor for Blood stream infection
  Groups: No of Positive CLABSI; Primary Blood stream infection; Secondary Blood stream infection

SUMMARY:
* Review key history and clinical examination findings of cases with CLABSI.
* Microbiological diagnosis and Culture sensitivity tests by automated Bact Alert and Vitek2c systems for CLABSI.
* Determine antibiotic biogram of each organism isolated
* Determine the prevalence of occurrence of Primary or secondary Blood stream infection, causing microorganism, and predisposing factors.

DETAILED DESCRIPTION:
Subjects and Methods

Study Design:

This cross-sectional descriptive study will be conducted on admitted patients in Cardiovascular Unit at the Tertiary Care Hospital in Port Said hospitals.

Subjects:

From each patient the following data will be collected: full medical history, symptoms and signs, lab investigations including serum electrolytes, procalcitonin, liver and kidney function tests, receipt of antibiotics and its response.

Inclusion criteria:

* Patients diagnosed with sepsis based on medical history, lab investigations and clinical picture.
* Both sex, and all age-groups.

Exclusion criteria:

* Patients diagnosed with sepsis proved by medical history, lab investigations and clinical picture who received non-beta lactam antibiotics for the past 24 hours.
* Samples proved contaminated by microbial flora will be rejected.

Methods:

Study design This study will be conducted at the tertiary care hospital which offers a medical and surgery ICU and also has a cardiovascular Unit.

Epidemiologic and clinical information of patients and classification of the bacteremia as Primary Bloodstream Infections (PBI), and Secondary Bloodstream Infections (SBI), based on CDC criteria (5) and its National Healthcare Safety Network (NHSN) yearly update.

Sample collection

1. Venous blood samples from cases with suspected sepsis, or bacteremia will be incubated with a medium which encourages promotes bacterial growth.
2. We will take samples of 2 or more sets of aerobic and anaerobic blood cultures (3or 8 mL per small or large bottle)
3. Two blood cultures drawn from different areas are frequently enough to diagnose bacteremia. Two out of 2 cultures growing identical type of bacteria often represents a real bacteremia, in particular if the organism which grows isn't a frequent contaminant.
4. Bacterial isolates from blood will be analysed by utilizing an automatic blood culture system (Bact/Alert).
5. Positive samples will be cultured on different selective media. Primary organism recognition will be done with matrix assisted laser desorption ionization time of flight MS on a Vitek MS system (BioMerieux, Inc. France).
6. Calibration will be performed using standard strains to validate the run.
7. Minimum Inhibitory Concentration (MIC) outcomes will be interpreted based on the Clinical and Laboratory Standards Institute (CLSI) protocols.
8. Biochemical tests which include CRP of Procalcitonin is most of time increased among cases with BSI.

Sample size:

Number of Samples is calculated according to the next equation:

N= (Z α\2)²×P(1-P)\d² (Daniel, 2009) In which; N= the required sample size (Z α\2) = A normal deviation reflect the type 1 error = 1.96 P = the prevalence of atypical bacteria in sputum samples = (46%) (13). D = the accuracy of estimate (how close to the true population) = 0.1

Thus; N= 60 blood samples.

Data Management and Statistical Analysis The results of the collected data will entered into SPSS-19 program for statistical analysis.

Descriptive data will be managed based on its type; mean, SD and range will summarize continuous data. While qualitative data will be summarized by frequencies.

With regard to analytic data, chi square test will be utilized to determine the difference between qualitative data, while T test and ANOVA will be utilized to determine the difference between quantitative data.

Ethical considerations

* The samples will be collected from patients after taking written informed consent.
* The study will be conducted after taking the permission from chairman of each department.
* The results of the patient will be confidential.
* The patient will be informed of the results and will be treated accordingly.
* The patient has the right to leave the study without compromising the patient's treatment or the patient's relationship with the care provider.

ELIGIBILITY:
Inclusion Criteria:

* • Patients diagnosed with sepsis based on medical history, lab investigations and clinical picture.

  * Both sex, and all age-groups.

Exclusion Criteria:

* Patients diagnosed with sepsis proved by medical history, lab investigations and clinical picture who received non-beta lactam antibiotics for the past 24 hours.

  * Samples proved contaminated by microbial flora will be rejected.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Venous blood samples from cases with suspected sepsis, or bacteremia will be incubated with a medium which encourages promotes bacterial growth.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
• Microbiological diagnosis and Culture sensitivity tests | 6 months
  • Microbiological diagnosis and Culture sensitivity tests by automated Bact Alert and Vitek2c systems for CLABSI.
Determine antibiotic biogram of each organism isolated | 6 months
  Determine antibiotic biogram of each organism isolated

SECONDARY OUTCOMES:
•Determine the prevalence of occurrence of Primary or secondary Blood stream infection | 4 months
  •Determine the prevalence of occurrence of Primary or secondary Blood stream infection, causing microorganism, and predisposing factors.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Prof. Refat Sadeq, Port Said
  - Faculty of Medicine Portsaid Uni, Port Said

IPD SHARING:
Plan to Share IPD: Yes
Publication in Medical journals
Supporting Information: CSR
Time Frame: after one year